CLINICAL TRIAL: NCT01798979
Title: A Phase I, Open Interaction Study Between Oral Doses of GLPG0634 (200 mg QD) and Single Oral Doses of Midazolam (2 mg) in Healthy Subjects
Brief Title: A Phase I, Open Interaction Study Between GLPG0634 and Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0634-CL-103
Record Dates: First submitted 2013-02-24; First posted 2013-02-26 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG0634; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Midazolam and GLPG0634 (Experimental): Each subject will receive a single oral dose of midazolam (2 mg) on 2 occasions (Days 1 and 8) and multiple oral doses of GLPG0634 (200 mg daily for 7 days) from Days 2 to 8.
  Interventions: Drug: GLPG0634; Drug: Midazolam

INTERVENTIONS:
Drug: GLPG0634 — Each subject will receive multiple oral doses of GLPG0634 (200 mg daily for 7 days) from Days 2 to 8.
Drug: Midazolam — Each subject will receive a single oral dose of midazolam (2 mg) on 2 occasions (Days 1 and 8)

SUMMARY:
This will be a drug-drug interaction study to evaluate the effect of multiple oral doses of GLPG0634 on the single dose pharmacokinetic profile of midazolam administered in fasted normal healthy males. Each subject will receive a single oral dose of midazolam (2 mg) on 2 occasions: on Day 1, before dosing with GLPG0634 and on Day 8, after multiple oral doses of GLPG0634 (daily for 7 days).

Also, the safety and tolerability of multiple oral doses of GLPG0634 co-administered with midazolam in healthy male subjects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* male, between 40 and 60 years of age, inclusive
* within BMI range 18 to 30 kg/m2, inclusive

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The amount of (1'-OH) Midazolam in plasma over time before and after multiple oral doses of GLPG0634 | Between predose and up to 24h postdose on Day 1 and Day 8
  To characterize the amount of (1'-OH) Midazolam in plasma over time before and after multiple doses of GLPG0634 - pharmacokinetics (PK) - in healthy subjects

SECONDARY OUTCOMES:
The amount of GLPG0634 and metabolite in plasma over time after multiple oral doses of GLPG0634 (and co-administration of Midazolam on Day 8) | Between predose (Day 2) and up to 96h after the last dose on Day 8 (on Day 12)
  To characterize the amount of GLPG0634 and metabolite in plasma over time after multiple doses of GLPG0634 (and co-administration of Midazolam on Day 8) - pharmacokinetics (PK) - in healthy subjects
Number of adverse events | Between screening and 7-10 days after the last dose of GLPG0634 (Day 15-18)
  To evaluate the safety and tolerability of GLPG0634 after multiple oral doses in healthy subjects with or without coadministration of Midazolam in terms of the number of adverse events reported
Changes in vital signs as measured by pulse, supine blood pressure, oral temperature (and respiratory rate only 1 hour post Midazolam dosing) | Between screening and 7-10 days after the last dose of GLPG0634 (Day 15-18)
  To evaluate the safety and tolerability of GLPG0634 after multiple oral doses in healthy subjects with or without coadministration of Midazolam in terms of changes in vital signs as measured by pulse, supine blood pressure, oral temperature (and respiratory rate) reported
Changes in 12-lead ECG measures | Between screening and 7-10 days after the last dose of GLPG0634 (Day 15-18)
  To evaluate the safety and tolerability of GLPG0634 after multiple oral doses in healthy subjects with or without coadministration of Midazolam in terms of changes in 12-ECG measures reported
Changes in physical exam measures | Between screening and 7-10 days after the last dose of GLPG0634 (Day 15-18)
  To evaluate the safety and tolerability of GLPG0634 after multiple oral doses in healthy subjects with or without coadministration of Midazolam in terms of changes in physical examination reported
Changes in blood safety lab parameters | Between screening and 7-10 days after the last dose of GLPG0634 (Day 15-18)
  To evaluate the safety and tolerability of GLPG0634 after multiple oral doses in healthy subjects with or without coadministration of Midazolam in terms of changes in blood safety lab parameters reported
Changes in urine safety lab parameters | Between screening and 7-10 days after the last dose of GLPG0634 (Day 15-18)
  To evaluate the safety and tolerability of GLPG0634 after multiple oral doses in healthy subjects with or without coadministration of Midazolam in terms of changes in urine safety lab parameters reported

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States